CLINICAL TRIAL: NCT04859166
Title: Prospective Primary Human Lungcancer Organoids to Predict Treatment Response
Acronym: Organoids lung
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Organoids lung
Record Dates: First submitted 2021-04-15; First posted 2021-04-26 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer
Keywords: Organoids; Lung; Cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Microphysiological Systems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A part of the tumor of approximately 1 cm3 will be removed from the primary tumor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Organoids — A part of the tumor of approximately 1 cm3 will be removed from the primary tumor.

SUMMARY:
Organoids are generated from tumor biopsies, taken during a standard procedure. and are a collection of organ-specific cell types that are able to self-organize in-vitro in a manner similar to the in-vivo situation (3D). They have the capability to facilitate in-depth analysis of patient's own tumor material at point of diagnosis and during progressive/recurrent disease. There is currently no published protocol to establish long-term lung cancer organoids from lung cancer patients. Such a methodology would enable the prospective identification of 'patient tailored optimal treatments" as well as the derivation of predictive biomarkers for response and relapse. Apart from organoids, xenograft models also still have their merits. To generate PDX, tumor material will be retrieved from surgical specimens, cut in small pieces, transplanted in the recipient immune deficient animals either subcutaneously or implanted directly into the lung. A tumor with the median growth rate will be serially transplanted in vivo for further therapeutic experiments. Dedicated small animal irradiaton in our facility enables precise local irradiation of lung tumors with minimal radiation exposure of the surrounding normal tissues. Integrated cone beam computed tomography imaging system allows longitudinal monitoring of tumor response to novel treatments.

DETAILED DESCRIPTION:
One of the most important barriers to achieve durable responses in advanced lung cancer is intra- and inter-tumor heterogeneity, a common feature of human solid cancers. Tumor heterogeneity is thought to be driven by a subpopulation of tumor cells termed lung cancer initiating cells or lung cancer stem cells that reflect the 'cell or origin" and maintain self-renewaland multipotent properties of these cells but that are transformed. Organoid technology has enabled the culturing of normal and transformed 'stem cells" directly from patients without any genetic manipulation (i.e.IPS). Such normal and cancer organoids maintain many of the properties of the tumors and are thought to be an excellent in vitro 3D model system. In a lab, investigators have successfully established primary 2D and 3D cell culture systems including organoids from the proximal bronchus coming from lobectomies. They are using these systems to predict normal tissue complication to combination treatments. It has been demonstrated that lung stem cell pathways such as the NOTCH signaling pathway are frequently deregulated in lung cancers and is associated with a worse outcome. In vitro and in preclinical models deregulation of the NOTCH pathway is associated with resistance to radiotherapy and first-line chemotherapy. Thus blocking the NOTCH pathway may improve treatment response. Checkpoint inhibitors have changed the outcome of patients with metastatic non-small cell lung cancer (NSCLC) in first and in second line, with improved progression-free survival (PFS), overall survival (OS) and quality of life. Radiotherapy has consistently been shown to activate key elements of the immune system that are responsible for resistance for immune therapy. Radiation upregulates MHC-class I molecules that many cancer cells lack or only poorly express, tumor-associated antigens, provokes immunogenic cell death, activates dendritic cells, decreases regulatory T-cells (Tregs) in the tumor, broadens the T-cell repertoire and increases T-cell trafficking, amongst many other effects. Radiation may convert a completely or partly poorly or non-immunogenic tumor immunogenic. Radiotherapy in combination with different forms of immune therapy such as anti-PD-(L)1, anti-CTLA4, immunocytokines, dendritic cell vaccination and Toll-like receptor agonists improved consistently local tumor control and very interestingly, lead to better systemic tumor control (the "abscopal" effect) and the induction of specific anti-cancer immunity with a memory effect. Moreover, as PD1/PD-L1 is upregulated by radiation and radiation can overcome resistance for PD-(L)1 blockage, their combination is logical. The best timing, sequencing and dosing of all modalities is a matter of intense research. Radiotherapy may well become an integral part of immune therapy against cancer. Nevertheless, as with all treatments, optimal biomarkers for response are lacking. They would not only allow patient selection, but would also give insight in resistance mechanisms and the identification of new targets or the optimal use of current medications and radiation, such as dosing and sequencing. Moreover, not only biomarkers for tumor response, but also for side effects are needed, for the latter may be dose-limiting and result in the omission of therapy in the more frail and older patient population. Putative biomarkers for immune response are those associated with immunogenic cell death (ICD). Organoids are generated from tissue biopsies, and are a collection of organ-specific cell types that are able to self-organize in-vitro in a manner similar to the in-vivo situation (3D). They have the capability to facilitate in-depth analysis of patient's own tumor material at point of diagnosis and during progressive/recurrent disease. There is currently no published protocol to establish long-term lung cancer organoids from lung cancer patients. Such a methodology would enable the prospective identification of 'patient tailored optimal treatments" as well as the derivation of predictive biomarkers for response and relapse. Apart from organoids, xenograft models also still have their merits. In xenografts, human tumor cells or pieces are injected in immunocompromised mice. Especially xenografts derived from fresh human cancer specimen have gained much attention for the same tumor as in an individual patient can be grown in a mice allowing to study the response to therapy and the mechanisms of resistance. Patient-derived tumor xenograft (PDX) models are more reflective of patient population in terms of the parental tumors' histomorphological characteristics, the effect of clonal selection and evolution on maintaining genomic integrity in low-passage PDXs compared to the donor tissue. While organoids can give many insights into molecular biology of the response to various anti-cancer therapies, in vivo models allow testing novel anti-cancer therapeutic approaches taking complex tumor microenvironment into account reflecting at least in part clinical situation. As a clinically representative tool that best recapitulates the biological properties of their respective tumor type, PDX models could serve as an important aid in personalized medicine studies as well. The tumor can be transplanted subcutaneously, but more recently also orthotopically (e.g. a breast cancer is transplanted in the breast of a mouse) to investigate the interaction between the tumor and the environment. In Maastro lab, we have experience with a variety of these models including orthotopic lung tumor models. To generate PDX, tumor material will be retrieved from surgical specimens, cut in small pieces, transplanted in the recipient immune deficient animals either subcutaneously or implanted directly into the lung. A tumor with the median growth rate will be serially transplanted in vivo for further therapeutic experiments. Dedicated small animal irradiator in the investigators facility enables precise local irradiation of lung tumors with minimal radiation exposure of the surrounding normal tissues. Integrated cone beam computed tomography imaging system allows longitudinal monitoring of tumor response to novel treatments.

ELIGIBILITY:
Inclusion Criteria:

- Undergo primary surgical resection of a primary lung cancer (e.g. wedge resection, segmental resection, lobectomy, pneumonectomy)

Exclusion Criteria:

- Preceding induction treatment (e.g. induction chemotherapy or chemo-radiotherapy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In a one year period,30 patients who are selected to undergo surgical removal of a primary lung cancer will be included. The tumor material that will be used to make organoids will be derived from 'left-over' tumor tissue that is not needed for the pathologist to make a diagnosis, to stage the patient or to perform a molecular diagnosis. The patient therefore does not require to undergo additional treatments or procedures.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Bio-banking | 5 years
  To establish long term culturing and bio-banking conditions for primary lung cancer organoids.
Frequency of organoid formation | 5 years
  To determine the frequency of primary, secondary and tertiary organoid formation
Distribution | 5 years
  The size distribution of the organoids
Proliferation | 5 years
  The rate of proliferation and cell death (turnover) will be calculated
PDX models of lung cancer | 5 years
  To establish PDX models of lung cancer by means of passaging and expansion through subcutaneous engraftment in immune deficient animals and create PDX tumor bank for subsequent experiments
Established PDX histologically | 5 years
  To characterize established PDX histologically and to compare these characteristics with donor tissue
Established PDX genetically | 5 years
  To characterize established PDX genetically (most frequently occurring driver mutations in lung cancer) and to compare these characteristics with donor tissue
Established PDX biologically | 5 years
  To characterize established PDX biologically (proliferation, tumor microenvironment, etc.) and to compare these characteristics with donor tissue
Test treatments | 5 years
  Using PDX models to test novel anti-cancer treatments such as a hypoxia-activated prodrug (HAP) in combination with radiation
Test treatments | 5 years
  Using PDX models to develop predictive assay of tumor response to HA

SECONDARY OUTCOMES:
Test hypotheses | 5 years
  The organoids will be used to test hypotheses such as epi-genetic stability, response to targeted and cytotoxic therapies
Generate cell lines | 5 years
  Use the PDX to generate cancer cell lines for in vitro assays to test intrinsic sensitivity of cells to HAPs and other drugs in 2D and 3D settings

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vooijs, MD, PhD, Principal Investigator — Maastro
Locations (2):
- Netherlands (2):
  - Zuyderland Medical Center, Heerlen
  - Maastro, Maastricht